CLINICAL TRIAL: NCT01919450
Title: Characterization of Myocardial Blood Flow Measurements Using Lexiscan®™ (Regadenoson) (Lexiscan®™) Rubidium-82 Myocardial Perfusion PET: A Temporal-Dependency Investigation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Timothy M. Bateman, MD (Industry)
Responsible Party: Sponsor-Investigator, Timothy M. Bateman, MD, Medical Director, Cardiovascular Imaging Technologies
Organization: Cardiovascular Imaging Technologies (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-058
Record Dates: First submitted 2013-07-25; First posted 2013-08-09 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Myocardial Blood Flow Reserve
Keywords: PET; Lexiscan; Regadenoson; Rubidium; Blood Flow Reserve; Myocardial Perfusion; Quantitated Myocardial Perfusion
MeSH Terms: interventions — regadenoson; Rubidium-82

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 10 Second Delay (Active Comparator): A 10 second delay is imposed between the Lexiscan (Regadenoson) injection and start of myocardial perfusion PET imaging.
  Interventions: Drug: Regadenoson; Radiation: Rubidium-82
- 2 Minute Delay (Active Comparator): A 2 minute delay is imposed between the Lexiscan (Regadenoson) injection and start of myocardial perfusion PET imaging.
  Interventions: Drug: Regadenoson; Radiation: Rubidium-82
- 4 Minute Delay (Active Comparator): A 4 minute delay is imposed between the Lexiscan (Regadenoson) injection and start of myocardial perfusion PET imaging.
  Interventions: Drug: Regadenoson; Radiation: Rubidium-82
- 1 Minute Delay (Active Comparator): A 1 minute delay is imposed between the Lexiscan (Regadenoson) injection and start of myocardial perfusion PET imaging.
  Interventions: Drug: Regadenoson; Radiation: Rubidium-82

INTERVENTIONS:
Drug: Regadenoson — Subjects will undergo a rest/Lexiscan (regadenoson) stress myocardial perfusion PET study.
  Other Names: Lexiscan
Radiation: Rubidium-82 — Subjects undergo a rest/Lexiscan (regadenoson) stress myocardial perfusion PET study.
  Other Names: Cardio-Gen82

SUMMARY:
The purpose of this study is to evaluate the consistency of quantitative peak stress myocardial blood flow and myocardial blood flow reserve following a 10 second, 1 minute, 2 minute or 4 minute delay in beginning the rubidium-82 infusion post-Lexiscan (regadenoson) injection. It is anticipated that there will be no or minimal difference between the four delay times.

ELIGIBILITY:
Inclusion Criteria:

* Recent normal clinically-indicated exercise myocardial perfusion SPECT, treadmill maximal exercise test or exercise echocardiographic study
* No change in symptoms between the exercise study and PET study
* Capable of providing written informed consent
* BMI 25-32 kg/m2

Exclusion Criteria:

* Diabetes mellitus
* Coronary Artery Calcium Score >25
* Second and Third Degree Atrioventricular Node Block
* Sinus Node Dysfunction
* Recent Syncope of unknown etiology
* Left ventricular hypertrophy per ECG or echocardiography
* Slowed circulation times
* Active wheezing or with acute asthmatic or bronchospastic attacks requiring changes in therapy within the past 30 days.
* Patients that have experienced a previous hypersensitivity reaction thought to be related to Lexiscan

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Bateman, MD, Principal Investigator — Cardiovascular Imaging Technologies
Locations (1):
- Saint Luke's Hospital Imaging Center, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with a low pretest likelihood for CAD based on gender, symptoms and recent (<90 days) normal-clinically-indicated TMET, exercise echocardiogram or exercise myocardial perfusion SPECT test were recruited for consent and participation.
Period: Overall Study
Arm/Group | 10 Second Delay | 2 Minute Delay | 4 Minute Delay | 1 Minute Delay
Started | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 19
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 Second Delay | 2 Minute Delay | 4 Minute Delay | 1 Minute Delay | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.5 (13.8) | 51.3 (10.4) | 53.1 (9.6) | 50.6 (9.9) | 51.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 10 | 15 | 45
  Male | 6 | 14 | 10 | 5 | 35
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: Measure Quantitated Myocardial Perfusion Reserve After a 4 Minute Delay in Lexiscan (Regadenoson)
Description: The end-point of this study is to establish the mean and standard deviations of myocardial blood flow reserve (peak stress to rest ratio) values based on a 10 second, 1 minute, 2 minute and 4 minute delays between Lexiscan (Regadenoson) injection and the start of myocardial perfusion PET imaging.
Time Frame: 4 minutes
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | 4 Minute Delay
Number analyzed (Participants) | 18
Ratio | 2.57 (0.71)

2. Primary Outcome: Measure Quantitated Myocardial Perfusion Reserve After a 2 Minute Delay in Lexiscan (Regadenoson)
Description: as for outcome 1
Time Frame: 2 mintues
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | 2 Minute Delay
Number analyzed (Participants) | 19
Ratio | 2.93 (0.7)

3. Primary Outcome: Measure Quantitated Myocardial Perfusion Reserve After a 10 Second Delay in Lexiscan (Regadenoson)
Description: as for outcome 1
Time Frame: 10 seconds
Measure: Median (Standard Deviation); unit: Ratio
Arm/Group | 10 Second Delay
Number analyzed (Participants) | 19
Ratio | 2.34 (.38)

4. Primary Outcome: Measure Quantitated Myocardial Perfusion Reserve After a 1 Minute Delay in Lexiscan (Regadenoson)
Description: as for outcome 1
Time Frame: 1 minute
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | 1 Minute Delay
Number analyzed (Participants) | 18
Ratio | 2.76 (.56)

ADVERSE EVENTS:
Time Frame: Adverse events were collected immediately post-informed consent and through the patient's entire visit to the imaging facility.
Description: AEs were recorded on an Adverse Event (AE) log. The AE log consisted of: 1.) Description of event; 2.) Start and stop time of event; 3.) Severity of event; 4.) Likelihood that the event was related to the study drug; 5.) Relationship of event to other test procedures; 6.) Any treatment actions taken, and 7.) the final outcome.
Arm/Group | 10 Second Delay | 2 Minute Delay | 4 Minute Delay | 1 Minute Delay
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 1/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 Second Delay (N=20) | 2 Minute Delay (N=20) | 4 Minute Delay (N=19) | 1 Minute Delay (N=20)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — 1 subject was admitted to ED 4 days post-study participation with chest/neck pain, predating study. Based upon symptoms and palpable left lateral neck discomfort, pt. was dismissed with a dx of musculoskeletal etiology.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No